CLINICAL TRIAL: NCT01235377
Title: Tolerance to Target Doses of Thiazides in Actual Practice: A Feasibility Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Pharmacy Benefits Management Strategic Healthcare Group (U.S. Federal Agency)
Responsible Party: Principal Investigator, Madeline McCarren, Biostatistician, VA Pharmacy Benefits Management Strategic Healthcare Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VMS156
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Results first posted 2014-11-25 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Hypertension
Keywords: prescribing patterns; thiazide; chlorthalidone; hydrochlorothiazide; target dose; cluster randomized trial
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Favor Chlorthalidone (Active Comparator): Providers randomized to Favor Chlorthalidone will have agreed to prescribe chlorthalidone for patients who are to be newly prescribed a thiazide for hypertension, whether the thiazide is 1st line or add-on therapy. This cluster designation applies only for patients for whom there is equipoise; providers are expected to deviate if medically indicated for individual patients
  Interventions: Other: Favor one of two thiazides for new prescriptions & attempt target dose
- Favor Hydrochlorothiazide (Active Comparator): Providers randomized to Favor Hydrochlorothiazide will have agreed to prescribe hydrochlorothiazide for patients who are to be newly prescribed a thiazide for hypertension, whether the thiazide is 1st line or add-on therapy. This cluster designation applies only for patients for whom there is equipoise; providers are expected to deviate if medically indicated for individual patients
  Interventions: Other: Favor one of two thiazides for new prescriptions & attempt target dose

INTERVENTIONS:
Other: Favor one of two thiazides for new prescriptions & attempt target dose — Providers will be randomized to either Favor Chlorthalidone or Favor Hydrochlorothiazide for patients who are to be newly prescribed a thiazide for hypertension, whether the thiazide is 1st line or add-on therapy. Providers will have agreed to adhere to their assignment for patients for whom there is equipoise, but they are free to deviate if medically indicated for individual patients. There is no requirement to maintain the initial thiazide therapy; it is expected that the regimen may require adjustment over time. The cluster assignment is simply to favor a particular thiazide on initiation of thiazide therapy and attempt to reach the target dose.

SUMMARY:
This is a pilot study of a method to compare common, FDA-approved drugs in a clinic. Instead of putting single patients into one of two drug groups, the investigators will assign the doctors who prescribe these drugs for high blood pressure into two groups. One group of doctors has agreed to prescribe mostly ("favor") one drug, chlorthalidone, if that drug would be a good choice for a patient. The other group has agreed to prescribe mostly hydrochlorothiazide. For both groups, they will try to use the doses that were shown to be protective in other trials. If the doctors mostly prescribe the drug they agreed to favor, the investigators will be able to compare outcomes, like heart attacks, in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* VA prescribers of thiazides for hypertension

Exclusion Criteria:

* at non-participating VA sites

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2013-10 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madeline McCarren, PhD, MPH, Principal Investigator — VA Pharmacy Benefits Management
Locations (5):
- United States (5):
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - Charles George VAMC, Asheville, North Carolina
  - Wilkes-Barre VA Medical Center, Wilkes-Barre, Pennsylvania
  - WJB Dorn VA Medical Center, Columbia, South Carolina
  - WJB Dorn VAMC/Columbia Orangeburg VA Outpatient Clinic, Orangeburg, South Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Favor Chlorthalidone: Providers randomized to Favor Chlorthalidone agreed to prescribe chlorthalidone for patients who are to be newly prescribed a thiazide for hypertension. This cluster designation applies only for patients for whom there is equipoise; providers are expected to deviate if medically indicated for individual patients
- Favor Hydrochlorothiazide: Providers randomized to Favor Hydrochlorothiazide agreed to prescribe hydrochlorothiazide for patients who are to be newly prescribed a thiazide for hypertension. This cluster designation applies only for patients for whom there is equipoise; providers are expected to deviate if medically indicated for individual patients
Period: Overall Study
Arm/Group | Favor Chlorthalidone | Favor Hydrochlorothiazide
Started | 11 | 9
Completed | 10 | 8
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: patients of the 18 providers
Groups:
- Total: Total of all reporting groups
Arm/Group | Favor Chlorthalidone | Favor Hydrochlorothiazide | Total
Number analyzed (Participants) | 77 | 61 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (10.8) | 60.4 (13.1) | 60.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 76 | 60 | 136

OUTCOME MEASURES:

1. Primary Outcome: Prescription Rates
Description: rates of provider prescribing of the Cluster Designated drug
Time Frame: nine months
Population: providers prescribing a thiazide at least once in the study period
Measure: Median (Inter-Quartile Range); unit: % new thiazide prescriptions
Arm/Group | Favor Chlorthalidone | Favor Hydrochlorothiazide
Number analyzed (Participants) | 10 | 8
% new thiazide prescriptions | 80 [54.5 to 100] | 100 [100 to 100]

2. Secondary Outcome: Factors Associated With Prescribing Patterns
Description: factors (barriers and facilitators) associated with prescribing according to the Cluster Designation
Time Frame: nine months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Favor Chlorthalidone | Favor Hydrochlorothiazide
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/61
Other Adverse Events (participants affected / at risk) | 2/77 | 0/61
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Favor Chlorthalidone (N=77) | Favor Hydrochlorothiazide (N=61)
other abnormal glucose (Endocrine disorders) | 2 | 0 — from analysis of select International Classification of Diseases (ICD9) terms in an administrative database

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes